CLINICAL TRIAL: NCT04118868
Title: Phase 1B, Pilot Study to Assess the Pharmacodynamics, Pharmacokinetics, Safety, Activity of Pembrolizumab Administered Intra-lymphatically Using the Sofusa® DoseConnect™ in Patients With Relapsed/Refractory Cutaneous T- Cell Lymphoma (CTCL)
Brief Title: Pembrolizumab Administered Via the Sofusa® DoseConnect™ in Patients With Relapsed/Refractory Cutaneous T-cell Lymphoma.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STI-SOFUSA-1001
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Mycosis Fungoides
Keywords: CTCL; Cutaneous T-cell Lymphoma; MF/SS; Mycosis Fungoides; pembrolizumab; PD-L1
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All participants (Experimental): Pembrolizumab administered intralymphatically using the Sofusa® DoseConnect™device
  Interventions: Combination Product: Pembrolizumab administered using the Sofusa® DoseConnect™

INTERVENTIONS:
Combination Product: Pembrolizumab administered using the Sofusa® DoseConnect™ — pembrolizumab will be administered intralymphatically using the Sofusa® DoseConnect™ device
  Other Names: Keytruda® administered using Sofusa® DoseConnect™ device

SUMMARY:
In this pilot study, pembrolizumab will be administered via DoseConnect in patient with relapsed or refractory cutaneous T-cell lymphoma to assess through pharmacodynamic assessment in the tumor tissue to assess if lymphatic delivery of pembrolizumab using Sofusa DoseConnect is feasible.

DETAILED DESCRIPTION:
This is an open-label, single-center pilot study to investigate the pharmacodynamics, pharmacokinetics (PK), safety, and activity of pembrolizumab administered intra-lymphatically using the DoseConnect in participants with relapsed or refractory cutaneous T-cell lymphoma (CTCL).

All participants will receive the study intervention, pembrolizumab administered intralymphatically using the Sofusa DoseConnect device.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of Mycosis fungoides (MF)
* Stage IB to IIIB disease at screening
* Received at least 1 previous line of systemic therapy for CTCL. (Participants with CD 30 positive MF must have received prior treatment with brentuximab vedotin.)
* Documented disease progression during or after the last therapy.
* Not previously treated with transplant and is ineligible for transplant
* Willing to undergo two biopsies during the study
* 18 years or older at the time of signing informed consent form (ICF)
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Females of childbearing potential (FCBP) must agree to use a reliable form of contraceptive for the duration of the study and for at least 120 days (4 months) following the last dose of study intervention.
* Male participants must agree to use barrier contraception (i.e., condoms) for the duration of the study and for at least 120 days (4 months) following the last dose of study intervention

Exclusion Criteria:

* Disease with extensive visceral or blood involvement.
* Previously treated with an anti-PD-L1 or anti-PD-1 antibody
* Any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo, hormone replacement therapy for stable thyroid diseases and Type 1 diabetes mellitus.
* Prior allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation.
* Known seropositive for or have active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV), or human immunodeficiency virus (HIV)
* History of interstitial lung disease
* History of severe hypersensitivity reactions to other monoclonal antibodies or known hypersensitivity to the study intervention or its excipients, indocyanine green dye or iodine.
* Known current drug or alcohol abuse.
* Pregnant or lactating.
* Underlying medical condition resulting in abnormally slow lymphatic flow as determined by the Investigator.
* Require immediate treatment for MF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-01-29 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic effect of pembrolizumab administered by the Sofusa® DoseConnect™ device | Approximately 14 months
  T-cell exhaustion/activation markers: PD-1, Lag-3, Tim-3, ICOS, HLA-DR and Granzyme B in CD3+CD4+ malignant and CD3+CD8+ tumor-infiltrating T-cells in tumor tissue

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of pembrolizumab administered by the Sofusa® DoseConnect™ device | Approximately 24 months
  Terms, frequency, severity and seriousness of adverse events (AEs) and relationship of AEs to pembrolizumab and/or Sofusa® DoseConnect™
Area Under the Curve (AUC) of the blood levels of pembrolizumab | Approximately 17 months
  Measure the actual body exposure to pembrolizumab
Maximum Plasma Concentration (Cmax) of pembrolizumab | Approximately 17 months
  Measure the maximum (or peak) blood concentration of pembrolizumab
Time of Maximum concentration observed (Tmax) of pembrolizumab | Approximately 17 months
  Measure the is the time at which the maximum blood concentration of pembrolizumab is observed
Half-life (t1/2) of pembrolizumab | Approximately 17 months
  Measure the time it takes for the concentration of the pembrolizumab in the blood to be reduced by 50%

CONTACTS AND LOCATIONS:
Overall Officials: Andreas G Niethammer, MD PhD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- City of Hope, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narducci MG, Tosi A, Frezzolini A, Scala E, Passarelli F, Bonmassar L, Monopoli A, Accetturi MP, Cantonetti M, Antonini Cappellini GC, De Galitiis F, Rosato A, Picozza M, Russo G, D'Atri S. Reduction of T Lymphoma Cells and Immunological Invigoration in a Patient Concurrently Affected by Melanoma and Sezary Syndrome Treated With Nivolumab. Front Immunol. 2020 Sep 25;11:579894. doi: 10.3389/fimmu.2020.579894. eCollection 2020. PMID 33072126